CLINICAL TRIAL: NCT04451109
Title: Dilapan-S®: A Multicenter US E-registry
Status: Active, not recruiting | Type: Observational
Sponsor: Medicem Technology s.r.o. (Other)
Collaborators: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: Dilapan-S US E-registry
Record Dates: First submitted 2020-06-17; First posted 2020-06-30 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Post Term Pregnancy; Premature Rupture of Membrane; Fetal Growth Retardation; Oligohydramnios; Gestational Diabetes; High Blood Pressure in Pregnancy
Keywords: induction of labour; induction of labor; labour induction; labor induction; Dilapan; dilator; cervical ripening; cervical priming; preinduction; pre-induction
MeSH Terms: conditions — Pregnancy, Prolonged; Fetal Membranes, Premature Rupture; Fetal Growth Retardation; Oligohydramnios; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cases in which Dilapan-S was used for cervical ripening.: Every participating site will select 50 cases of pregnant women who underwent cervical ripening by Dilapan-S prior to induction of labor. These cases has to fulfill inclusion/exclusion criteria defined in the protocol.
  Interventions: Device: Dilapan-S

INTERVENTIONS:
Device: Dilapan-S — Application of Dilapan-S and all other procedures regarding cervical ripening and induction of labor will be carried out as per the hospital's standard practice.

SUMMARY:
Objective of this registry is to collect a representative set of real world data on the use of Dilapan-S® for pre-induction cervical ripening in daily clinical practice. Upon completion of the registry, relevant collected data will be analyzed and published.

DETAILED DESCRIPTION:
In the US, 23% of pregnant women undergo labor induction. A recent randomized controlled trial showed that elective labor induction at term in low-risk nulliparous women is associated with a lower risk of cesarean delivery and preeclampsia, with no increase in adverse perinatal morbidities. Hence, one can assume that labor induction rates will increase. The majority of women undergoing induction have unfavorable cervixes and require cervical ripening agents. Dilapan-S®, a hygroscopic cervical dilator made from a patented hydrogel (AQUACRYL), has been used in the past for cervical ripening for early gestation uterine evacuation. Dilapan-S® was approved by the FDA for cervical ripening in the third trimester in 2015.

The Dilapan-S® rods are inserted into the cervical canal, are contained within the vagina, and do not require tension. Dilapan-S® works by absorbing fluid from cervical canal cells, resulting in reversible cell membrane dehydration and softening. In addition, the increase in the rod's volume creates a mechanical stretch and leads to the release of endogenous prostaglandins, causing cervical ripening. Recently, a multicenter prospective cohort study showed that Dilapan-S® is a safe and effective method for cervical ripening in term gestations. Lastly, our group performed non-inferiority randomized clinical trial comparing Dilapan-S® to Foley balloon for cervical ripening in term pregnancies and found that Dilapan-S® is non-inferior to Foley balloon for pre-induction cervical ripening at term.

The Dilapan-S® rods are inserted into the cervical canal, are contained within the vagina, and do not require tension. Dilapan-S® works by absorbing fluid from cervical canal cells, resulting in reversible cell membrane dehydration and softening. In addition, the increase in the rod's volume creates a mechanical stretch and leads to the release of endogenous prostaglandins, causing cervical ripening. Advantages of Dilapan-S® over Foley include FDA approval, safe profile, no protrusion from the introitus, no need to keep under tension and better patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman whose plan of care is induction of labor
* Maternal age ≥ 18 years
* Gestational age ≥ 37 +0/7 weeks
* Dilapan-S® used for cervical ripening

Exclusion Criteria:

* Data not available for extraction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Selected patients fulfilling eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of overall vaginal delivery | right after child delivery

SECONDARY OUTCOMES:
Rate of vaginal delivery within 24 hours | 24 hours
Rate of vaginal delivery within 36 hours | 36 hours
Time to reach active stage of labor defined as ≥6 cm | 48 hours
  minutes
Change in Bishop score | 48 hours
  scale 0-13 (positive gain in Bishop score is considered to be a positive consequence of the intervention)
Rate of spontaneous vaginal delivery | right after child delivery
Rate of operative vaginal delivery | right after child delivery
Rate of caesarean sections | right after child delivery

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Saad, MD, Principal Investigator — The University of Texas Medical Branch, Galveston
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin JA, Hamilton BE, Osterman MJ, Driscoll AK, Mathews TJ. Births: Final Data for 2015. Natl Vital Stat Rep. 2017 Jan;66(1):1. PMID 28135188
- [Background] Grobman WA, Rice MM, Reddy UM, Tita ATN, Silver RM, Mallett G, Hill K, Thom EA, El-Sayed YY, Perez-Delboy A, Rouse DJ, Saade GR, Boggess KA, Chauhan SP, Iams JD, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Labor Induction versus Expectant Management in Low-Risk Nulliparous Women. N Engl J Med. 2018 Aug 9;379(6):513-523. doi: 10.1056/NEJMoa1800566. PMID 30089070
- [Background] Rayburn WF. Preinduction cervical ripening: basis and methods of current practice. Obstet Gynecol Surv. 2002 Oct;57(10):683-92. doi: 10.1097/00006254-200210000-00022. PMID 12368596
- [Background] Gupta J, Chodankar R, Baev O, Bahlmann F, Brega E, Gala A, Hellmeyer L, Hruban L, Maier J, Mehta P, Murthy A, Ritter M, Saad A, Shmakov R, Suneja A, Zahumensky J, Gdovinova D. Synthetic osmotic dilators in the induction of labour-An international multicentre observational study. Eur J Obstet Gynecol Reprod Biol. 2018 Oct;229:70-75. doi: 10.1016/j.ejogrb.2018.08.004. Epub 2018 Aug 3. PMID 30107363
- [Background] Saad AF, Villarreal J, Eid J, Spencer N, Ellis V, Hankins GD, Saade GR. A randomized controlled trial of Dilapan-S vs Foley balloon for preinduction cervical ripening (DILAFOL trial). Am J Obstet Gynecol. 2019 Mar;220(3):275.e1-275.e9. doi: 10.1016/j.ajog.2019.01.008. Epub 2019 Feb 18. PMID 30790569